CLINICAL TRIAL: NCT07055685
Title: Effects of Upper Limb Progressive Resistance Training Along With Core Stability Exercises on Pain, Core Strength and Upper Limb Balance in Cricket Fast Bowlers With Shoulder Injury
Brief Title: Effects of Upper Limb PRT With CSE on Pain, Core Strength and ULB in Cricket Fast Bowlers With Shoulder Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/828
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Resistance Training + Core Stability Exercises (Experimental)
  Interventions: Combination Product: Progressive Resistance Training + Core Stability Exercises
- Progressive Resistance Training (Experimental)
  Interventions: Combination Product: Progressive Resistance Training

INTERVENTIONS:
Combination Product: Progressive Resistance Training + Core Stability Exercises — Participants in Group A will engage in a combined program focusing on upper limb strengthening and trunk stabilization. The core stability component aims to improve neuromuscular control and trunk endurance, while the resistance training targets upper limb muscle strength and shoulder stability.
  Core Stability Exercises:
  Exercise Description Duration/Repetitions Planks Holding a straight-body position on elbows and toes. 30-60 seconds Bird-Dog Extending one arm and opposite leg, maintaining neutral spine. 5-10 sec/rep, 10-12 reps per side Dead Bug Supine position, extending opposite arm and leg. 3-5 sec/rep, 12-15 reps Bridging Lifting hips off ground, maintaining spinal alignment. 10-15 sec/rep, 12-15 reps Swiss Ball Stability Balance in sitting or leg lift positions using a Swiss ball. 20-30 sec/position, 10-12 reps Progression in core exercises will occur by increasing repetitions, duration, or complexity based on individual capability.
  Arms: Progressive Resistance Training + Core Stability Exercises
Combination Product: Progressive Resistance Training — will perform only the upper limb progressive resistance training protocol as outlined below. This regimen focuses on strengthening the shoulder complex, upper back, and arm muscles to improve muscular performance, endurance, and control. Progressive Resistance Training
  Arms: Progressive Resistance Training

SUMMARY:
Musculoskeletal pain and dysfunction, particularly in the upper limb and spine, are often linked to poor core stability and muscular imbalance. While progressive resistance training is a well-established approach to improve muscular strength, incorporating core stability exercises may provide additional benefits in terms of balance, posture, and neuromuscular control. However, limited studies have examined the combined effects of resistance and core stability training on upper limb strength, core endurance, pain reduction, and balance performance.

ELIGIBILITY:
Inclusion Criteria:

* Male cricket fast bowlers aged between 18 and 35 years.
* Diagnosed with shoulder injury (e.g., rotator cuff strain, impingement syndrome) confirmed by clinical assessment.
* History of shoulder pain for at least 4 weeks but not more than 6 months.
* Currently active in training or playing at club, district, or national level.(25)

Exclusion Criteria:

* History of shoulder surgery or dislocation within the past 1 year.
* Presence of neurological disorders or systemic conditions affecting shoulder function.
* Current participation in any other shoulder rehabilitation or strength training program.
* Structural deformities or congenital abnormalities of the upper limb.(26)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | 12 Months
  The Visual Analog Scale is a simple and validated tool widely used for the assessment of subjective pain intensity. It consists of a 10-centimeter horizontal line, with the endpoints defining the extremes of pain-'no pain' on the left end (0) and 'worst imaginable pain' on the right end . Participants mark a point on the line that corresponds to their perceived pain intensity. The distance in centimeters from the "no pain" end to the mark is measured to quantify pain. The VAS is sensitive to changes in pain and has high reliability and validity in both clinical and sports injury populations
Shoulder Pain and Disability Index (SPADI) | 12 Months
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire used to assess pain and functional disability in individuals with shoulder pathology. It consists of 13 items divided into two subscales: pain (5 items) and disability (8 items), each rated on a scale from 0 (no pain/difficulty) to 10 (worst pain/inability). SPADI has demonstrated excellent validity, with strong correlations to other functional assessment tools, and reliability, with high internal consistency (Cronbach's alpha 0.86-0.95) and test-retest reliability (ICC 0.89-0.93). Its responsiveness to clinical change makes it a valuable tool for both research and rehabilitation monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore City, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No